CLINICAL TRIAL: NCT02922309
Title: Voice Therapy for Benign Voice Disorders in the Elderly: A Randomized Controlled Trial Comparing Telepractice and Conventional Face-to-face Therapy
Brief Title: Comparing Telepractice and Conventional Face-to-face Voice Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chi-Te Wang, Attending Physician, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEMH-IRB-104193-E
Record Dates: First submitted 2016-09-23; First posted 2016-10-04 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Dysphonia; Aged; Speech Therapy
MeSH Terms: conditions — Dysphonia; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental (Experimental): Vocal Training via Telepractice
  Interventions: Behavioral: Vocal Training Via Telepractice
- control (Active Comparator): Vocal Training via face-to-face practice
  Interventions: Behavioral: Vocal Training Via face-to face practice

INTERVENTIONS:
Behavioral: Vocal Training Via Telepractice — Vocal Training Via Telepractice, delivered by integrated communication service
  Arms: experimental
Behavioral: Vocal Training Via face-to face practice — Vocal Training Via face-to face practice at medical facilities
  Arms: control

SUMMARY:
People over 55 years are high-risk with voice disorders. Voice disordered elderly need vocal training in order to improve communication efficiency and quality of life. However, participation in vocal training of elderly is often restricted by motivation, time of practice, and availability to hospital, which thus reduces treatment effects. The purpose of the study is to design a telecommunication vocal training system and a vocal training program for voice disordered elderly in Taiwan. The investigator proposed a 3-year consecutive study, including a single-blind, randomized controlled trial, to test the hypothesis that vocal training via telepractice for voice disordered elderly are not inferior to the standard face to face training.

DETAILED DESCRIPTION:
Randomization: per mutated block, 40 patients on each arms (experimental and control)

Allocation: sealed envelope indicating either of the 2 groups

Intervention: weekly vocal training, each course last for 30-40 minutes,lasting for 2 months

Outcome measurement: before treatment, 1 month, 3 months, and 6 months after treatment

Primary outcome: 10-item voice handicap index

Secondary outcome: acoustics and aerodynamic parameter

ELIGIBILITY:
Inclusion criteria:

* patient equal or older than 55 years old
* Voice Handicap Index-10 (VHI-10) score >10 point
* accessibility to a network connection

Exclusion criteria

* neurologic disorders
* active pulomanory disease
* mental disorder

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of 10-item voice handicap index at 2 months | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  min: 0(best); Max: 40(worst);

OTHER OUTCOMES:
Perceptual Analysis using grade, roughness, breathiness, asthenia, and strain | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  from 0(best) to 3(worst)
Jitter | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  percentage of jitter based on continuous vowel
Shimmer | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  decibel (dB) of shimmer based on continuous vowel
Noise to harmonic ratio | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  Noise to harmonic ratio based on continuous vowel
smoothed Cepstrum peak prominence | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  based on reading a Mandarin passage
Maximal phonation time | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  seconds
VLS | before treatment (after signing informed consent, prior to randomization) and within 2 weeks after the completion of voice therapy
  Videolaryngostroboscopy (mucosal wave: normal, mildly decreased, severely decreased, absent)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Te Wang, MD, PhD, Principal Investigator — Department of Otolaryngology, Far Eastern Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin FC, Chien HY, Chen SH, Kao YC, Cheng PW, Wang CT. Voice Therapy for Benign Voice Disorders in the Elderly: A Randomized Controlled Trial Comparing Telepractice and Conventional Face-to-Face Therapy. J Speech Lang Hear Res. 2020 Jul 20;63(7):2132-2140. doi: 10.1044/2020_JSLHR-19-00364. Epub 2020 Jun 24. PMID 32579859